CLINICAL TRIAL: NCT04415008
Title: A Prospective, Multicenter, Single Arm Clinical Study to Evaluate Efficacy of HAD Induction With Intensified Cytarabine in Newly-diagnosed CEBPA Double Mutated Acute Myeloid Leukemia
Brief Title: Efficacy of HAD Induction With Intensified Cytarabine in Newly-diagnosed CEBPA Double Mutated Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020008
Record Dates: First submitted 2020-05-31; First posted 2020-06-04 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: CEBPA Double Mutation; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental): prospective, open-label, multicenter,single arm
  Interventions: Drug: HAD induction with intermediate dose cytarabine

INTERVENTIONS:
Drug: HAD induction with intermediate dose cytarabine — daunorubicin,cytarabine,homoharringtonine

SUMMARY:
Acute myeloid leukemia is a heterogenous hematological malignancy, characterized by different cytogenetic or molecular features. CEBPA double mutation acute myeloid leukemia （CEBPAdm AML）has favourite prognosis, especially in younger adult patients. But cumulative incidence of relapse of this group patients is still high, so the treatment options need to be optimized urgently.HAD(homoharringtonine(HHT)+cytarabine+daunorubicin) with intermediate dose cytarabine improved the survival of AML, especially in patients with CEBPA double mutation.

DETAILED DESCRIPTION:
In this phase 2 study, 40 patients will be enrolled and treated with HAD induction regimen. High dose cytarabine will be given after complete remission achieved. The primary endpoint was event-free and relapse-free survival. Genetic mutations and measurable residual disease (MRD) will be detected at diagnosis and after chemotherapy. The risk stratification according to genetic mutations and MRD will also be explored.

induction chemotherapy:HHT 2mg/m2/d,day 1-7 cytarabine 100mg/m2/d, day1-4；1g/m2 /q12h ，day5-7 DNR 40mg/m2/d，day 1-3 re-induction chemotherapy:IDA 10mg/m2，day 1-3 cytarabine 100mg/m2，day 1-7 CTX 350mg/m2，day 2，day 5 consolidation chemotherapy: high dose cytarabine 3g/m2/Q12h,day1-3,for three cycles

ELIGIBILITY:
Inclusion Criteria:

* newly-diagnosed of acute myeloid leukemia except acute promyelocytic leukemia
* with CEBPA double mutation
* age≥ 14 years and<55 years，male or female
* ECOG-PS score 0-2
* laboratory tests（within 7 days before chemotherapy）

  1. serum total bilirubin≤1.5xULN；
  2. serum AST and ALT≤2.5xULN
  3. serum creatinine≤2xULN；
  4. cardiac enzymes≤2xULN
  5. ejection fraction >50% by ECHO。
* written informed consent。

Exclusion Criteria:

* subject has received remission induction chemotherapy
* secondary AML
* with other hematological malignancy
* with other tumors(needing treatment)
* pregnant or lactating women
* active heart diseases
* severe active infection
* unfit for enrollment evaluated by investigator

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 61 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-10-03 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
event free survival | 5 years
  Measured from day 1 of randomization to the date of treatment failure, hematologic relapse from CR or death from any cause, whichever occurs first
relapse free survival | 5 years
  survival from complete remission to relapse

SECONDARY OUTCOMES:
complete remission rate | 2.5 years
  incidence of complete remission after induction chemotherapy
early mortality | 2.5 years
  death during 30 days from induction chemotherapy
overall survival | 5 years
  duration from enrollment to death or loss of followup
RFS cencored at stem cell transplantation | 5 years
  RFS cencored at the date of stem cell transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- HBDH, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No